CLINICAL TRIAL: NCT03866590
Title: Pyruvate Kinase Deficiency Epidemiological Study. An International, Multicentre, Epidemiological Observational Study
Brief Title: Pyruvate Kinase Deficiency Epidemiological Study (PIECE)
Acronym: PIECE
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: PIECE 01-2019
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Pyruvate Kinase Deficiency
Keywords: Pyruvate Kinase Deficiency; Chronic anaemia; Biomarker
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients being at risk for Pyruvate Kinase Deficiency: Patients, older than 5 years and younger than 30 years old, being at risk for Pyruvate Kinase Deficiency, due to chronic anaemia or cholelithiasis or cholecystitis of undetermined aetiology

SUMMARY:
Pyruvate kinase deficiency (PKD) is the most common red cell glycolytic enzyme defect causing hereditary non-spherocytic hemolytic anemia, caused by mutations in the PKLR gene. The main goal of this study is the diagnosis of pyruvate kinase deficiency in patients who exhibit chronic anaemia and/or splenomegaly and/or judiance and/or hyperbilirubinemia and/or history of prolonged neonatal jaundice and/ or cholelithiasis of undetermined aetiology.

DETAILED DESCRIPTION:
Pyruvate kinase deficiency is the most common red cell glycolytic enzyme defect causing hereditary non-spherocytic hemolytic anemia, caused by mutations in the PKLR gene. PKLR encodes a pyruvate kinase that catalyzes the transphosphorylation of phosphoenolpyruvate into pyruvate and ATP. The current treatment options are red cell transfusions, chelation and splenectomy.

This is an international, multicentre, epidemiological and observational study.

The patients fulfilling the inclusion criteria will be enrolled into the Study and genetically tested for PKLR mutations via Next generation sequencing (NGS). Any mutation being detected by NGS, will be confirmed by Sanger sequencing.

PKLR-positive samples (homozygous or compound heterozygous for pathogenic variants) will be analysed for the identification of potential biomarkers via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared to a merged control samples in order establish a PKD specific biomarker.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent is obtained from the participant or legal representative
* The participant is equal or older than 5 years or equal or younger than 30 years old
* The participant exhibits the following symptoms of no obvious etiology:
* chronic anaemia and/or
* splenomegaly and/or
* jaundice and/or
* cholelithiasis and/or
* cholecystitis and/or
* hyperbilirubinemia and/or
* history of prolonged neonatal jaundice
* The participant is clinically diagnosed with PK deficiency

EXCLUSION CRITERIA:

* Inability to provide informed consent
* The participant does not suffer from chronic anaemia and splenomegaly and jaundice and cholelithiasis and cholecystitis and hyperbilirubinemia and history of prolonged neonatal jaundice
* The etiology of chronic anaemia or splenomegaly or jaundice or cholelithiasis or cholecystitis or kernicterus is clearly determined and is not due to PK deficiency
* The participant is younger than 5 years or older than 30 years old
* Previously enrolled in the PIECE Study
* Participant in custody

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients older than 5 years and younger than 30 years old, with high suspicion of PK deficiency, due to chronic anaemia or cholelithiasis or cholecystitis of undetermined aetiology
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Identification of 100 PKLR positive participants out of a cohort of 16,000 PK deficiency-suspected cases | 24 months
  Number of identified pyruvate kinase deficiency patients, which showing a mutation/pathogenic variant in their PKLR gene, within a cohort of 16.000 suspected cases via using respective patients' dry blood sample for confirmatory testing (next generation sequencing of PKLR gene)

SECONDARY OUTCOMES:
Biomarker/s establishment in PKLR-positive cohort | 24 months
  The quantitative determination of small molecules within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry, and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, M.D., Study Chair — CENTOGENE GmbH
Locations (1):
- Intervent Clinical Research Center, Pembroke Pines, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The plan will be defined at a later stages

REFERENCES:
- [Background] Beutler E, Gelbart T. Estimating the prevalence of pyruvate kinase deficiency from the gene frequency in the general white population. Blood. 2000 Jun 1;95(11):3585-8. PMID 10828047
- [Background] Grace RF, Bianchi P, van Beers EJ, Eber SW, Glader B, Yaish HM, Despotovic JM, Rothman JA, Sharma M, McNaull MM, Fermo E, Lezon-Geyda K, Morton DH, Neufeld EJ, Chonat S, Kollmar N, Knoll CM, Kuo K, Kwiatkowski JL, Pospisilova D, Pastore YD, Thompson AA, Newburger PE, Ravindranath Y, Wang WC, Wlodarski MW, Wang H, Holzhauer S, Breakey VR, Kunz J, Sheth S, Rose MJ, Bradeen HA, Neu N, Guo D, Al-Sayegh H, London WB, Gallagher PG, Zanella A, Barcellini W. Clinical spectrum of pyruvate kinase deficiency: data from the Pyruvate Kinase Deficiency Natural History Study. Blood. 2018 May 17;131(20):2183-2192. doi: 10.1182/blood-2017-10-810796. Epub 2018 Mar 16. PMID 29549173
- [Background] Carey PJ, Chandler J, Hendrick A, Reid MM, Saunders PW, Tinegate H, Taylor PR, West N. Prevalence of pyruvate kinase deficiency in northern European population in the north of England. Northern Region Haematologists Group. Blood. 2000 Dec 1;96(12):4005-6. No abstract available. PMID 11186276